CLINICAL TRIAL: NCT03696238
Title: Randomized, Parallel, Double-blind, Placebo Controlled, Study in Men to Assess the Influence of Aronox on Parameters Associated With Recovery Following Muscle Damaging Exercise
Brief Title: To Assess the Influence of Aronox on Parameters Associated With Recovery Following Muscle Damaging Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Givaudan France Naturals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NUAR01
Record Dates: First submitted 2018-09-25; First posted 2018-10-04 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2018-09

CONDITIONS: Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500mg of Aronox® >40% polyphenol aronia extract (Experimental): Name: Aronia PE 40% polyphenols Description: Powdered extract obtained from aronia berries (Aronia melanocarpa) Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg aronia extract Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX / Virage sante
  Interventions: Dietary Supplement: 500mg of Aronox® >40% polyphenol aronia extract
- 500mg of placebo (Placebo Comparator): Name: Placebo Description: Identical formulation as the treatment consisting of colored maltodextrin using artificial colors Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg placebo Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX (Advance nutraceutical) / Virage sante
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 500mg of Aronox® >40% polyphenol aronia extract — Name: Aronia PE 40% polyphenols Description: Powdered extract obtained from aronia berries (Aronia melanocarpa) Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg aronia extract Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX / Virage sante
  Arms: 500mg of Aronox® >40% polyphenol aronia extract
Other: Placebo — Name: Placebo Description: Identical formulation as the treatment consisting of colored maltodextrin using artificial colors Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg placebo Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX (Advance nutraceutical) / Virage sante
  Arms: 500mg of placebo

SUMMARY:
A randomized, double blind, counterbalanced, placebo controlled independent groups design. Prior to the visit, participants will be given a participant information sheet to inform of the procedure and requirements and undergo initial screening via email or telephone to ascertain suitability to participate. Stature, body mass, blood pressure and heart rate will be assessed. Participants will then be familiarized with the performance tests (MVC, vertical jump and sprint performance) and randomized to an investigational product group (2 groups: Aronox vs placebo; 1:1 allocation). The first investigational dose will be administered in the laboratory and participants will be given a 4-week supply of the investigational product to take in the morning with breakfast. Participants will also be asked to keep a food and activity diary for the 3 days preceding the baseline visit and for the duration of the damaging-recovery protocol.

Following this supplementation period (28 days), participants will be asked to return to the lab in a fed (not less than 2 hours prior to the visit) and hydrated state. Participants will also be asked to abstain from strenuous exercise and caffeine for 24 h prior to each lab visit. Stature, body mass, blood pressure and heart rate will be assessed. This will be followed by baseline assessment of muscle damage which will consist of visual analogue scales to assess lower limb muscle soreness (DOMS); pain pressure threshold and baseline measures of functional performance (maximal voluntary contraction, vertical jump performance and sprint performance) and limb girth. Furthermore, a blood sample will be taken to analyze creatine kinase (index of muscle damage). This will be followed by a strenuous bout of exercise designed to cause muscle damage comprising of 100 drop jumps from a 0.6 m platform at a rate of 1 jump every 10 seconds. A short rest will be provided after every 20 jumps. Each jump is performed by the participant stepping from the platform and landing two-footed on the floor and descending quickly to ~90° and 'explosively jumping upward with maximum effort. This model for muscle damage has been used on numerous occasions in the literature and has been used with great success in our own laboratory. Participants will then return to the lab at 24, 48 and 72 h post damaging protocol where muscle damage measures will be repeated to assess the level of recovery between the groups.

DETAILED DESCRIPTION:
A randomized, double blind, counterbalanced, placebo controlled independent groups design. Prior to the visit, participants will be given a participant information sheet to inform of the procedure and requirements and undergo initial screening via email or telephone to ascertain suitability to participate. If interested parties wish to participate, then they will be invited for a familiarisation visit, where they will:

* Be provided with an overview of the protocol and given the opportunity to ask questions
* Complete a health and physical activity questionnaire to ascertain study suitability
* Complete a training status questionnaire
* Assessment of ability to swallow capsules
* Complete an informed consent to participate in the study (assuming they meet the criteria and are willing to participate)

Stature, body mass, blood pressure and heart rate will be assessed. Participants will then be familiarized with the performance tests (MVC, vertical jump and sprint performance) and randomized to an investigational product group (2 groups: Aronox vs placebo; 1:1 allocation). The first investigational dose will be administered in the laboratory and participants will be given a 4-week supply of the investigational product to take in the morning with breakfast. Participants will also be asked to keep a food and activity diary for the 3 days preceding the baseline visit and for the duration of the damaging-recovery protocol.

Following this supplementation period (28 days), participants will be asked to return to the lab in a fed (not less than 2 hours prior to the visit) and hydrated state. Participants will also be asked to abstain from strenuous exercise and caffeine for 24 h prior to each lab visit. Stature, body mass, blood pressure and heart rate will be assessed. This will be followed by baseline assessment of muscle damage which will consist of visual analogue scales to assess lower limb muscle soreness (DOMS); pain pressure threshold and baseline measures of functional performance (maximal voluntary contraction, vertical jump performance and sprint performance) and limb girth. Furthermore, a blood sample will be taken to analyze creatine kinase (index of muscle damage). This will be followed by a strenuous bout of exercise designed to cause muscle damage comprising of 100 drop jumps from a 0.6 m platform at a rate of 1 jump every 10 seconds. A short rest will be provided after every 20 jumps. Each jump is performed by the participant stepping from the platform and landing two-footed on the floor and descending quickly to ~90° and 'explosively jumping upward with maximum effort. This model for muscle damage has been used on numerous occasions in the literature and has been used with great success in our own laboratory. Participants will then return to the lab at 24, 48 and 72 h post damaging protocol where muscle damage measures will be repeated to assess the level of recovery between the groups.

Exercise protocol details Muscle damage will be induced using a drop jump protocol our laboratory has used previously. It consists of 100 drop jumps performed 10 seconds apart with a 2-minute rest period provided every 20 jumps. Each jump will be conducted from a 0.6 m high box; upon landing, participants descend to a ~90º knee angle before performing a maximal effort vertical jump.

Passive muscle soreness will be reported on a 200 mm visual analogue scale and muscle site-specific soreness will be assessed as pressure pain threshold (PPT) with a handheld algometer (N2). Measurements were taken with participants lying supine; pressure was applied continuously at a rate of ~10 N cm-2∙s-1 until a pressure of ~40 N cm-2∙s-1 is achieved on the muscle belly; whereupon the participant will report muscle soreness on the aforementioned visual analogue scale.

Limb girth will be measured at the mid-thigh to examine limb swelling. This will be determined by identifying the midpoint between the inguinal crease and the superior border of the patella the right leg whilst the participant remained standing in anatomical zero. The location will be marked with permanent marker to ensure consistency on subsequent days.

A venous blood sample will then taken to examine creatine kinase (CK) concentrations to provide evidence that muscle damage has occurred.

Maximal isometric voluntary contractions (MIVCs) performed using a portable strain gauge (MIE Medical Research Ltd., Leeds, UK), will be used to examine strength loss and recovery. The peak value from 3 maximal contractions (separated by 60 seconds) will be used for analysis. In addition, counter movement jumps (CMJ) will be examined with an optical system to measure jump height in cm. With hands on their hips, participants will descend into a ~90° squat and jump vertically with maximal effort. The average of 3 maximal jumps (separated by 30 seconds) will be used for analysis. Participants will complete a single maximal effort 30 m sprint where sprint time will be recorded. The sprint will be initiated from a line 30 cm behind the start line in order to prevent false triggering of the timing gates (Brower, Utah, USA). In addition to the aforementioned measures that will be repeated at 24, 48 and 72 h, a perceived recovery questionnaire to assess more qualitative aspects of the intervention on recovery from the damaging protocol will be completed.

Supplementation and dietary control Following group allocation, participants will be provided with aronia (Aronox® ) or placebo (PLA) supplementation and instructed to consume 500mg of the investigational product. The PLA will consist of 95% maltodextrin with 5% artificial dyes (red lake and blue lake). The 500mg of Aronox is fortified with maltodextrin in order to provide 200 mg of polyphenol in total. Aronia consumption has shown no safety issues when used as an ingredient in dietary supplements or as a study drug in clinical trials by adults at dose levels ranging from 150 to 300 mg of extract per day for 14 days up to 2 months (Broncel et al., 2010; Naruszewicz et al., 2007).

Participants will be instructed not to consume the supplement on the day of initial assessment and consume the supplement after each laboratory visit as previous research (Bitsch et al. 2004; Kurilich et al. 2005) has demonstrated that systemic anthocyanin bioavailability increases to a peak between 1-2 hours post-ingestion. In addition, training logs will be kept to examine differences in training volume between groups and also general health log to record illness or consumption of any pharma during the supplementation period.

Data analysis

All data will be expressed as means ± SD, and statistical significance will be set at P < 0.05 prior to analyses. Differences in participant group characteristics, training history, and dietary intake were analysed using Student t-tests. Nutritics dietary analysis software (Nutritics LTD, Dublin, Ireland) will be used to analyse participant's food diaries. Dependent variables (MIVC, CMJ, VAS, and all blood indices) will be analysed using a mixed model ANOVA with 2 independent group levels (Aronex vs. PLA) and 4 repeated measures time points (pre, 24,48,72 h). If the ANOVA indicates a significant interaction effect (drink × time), Fisher LSD post hoc analysis will be performed to locate the significant differences. Homogeneity of variance will be checked with Mauchly's test of sphericity, and in the event of a significant result, GreenhouseGeisser adjustments will be used. All data will be analysed using IBM SPSS Statistics 22 for Windows (Surrey, UK).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men 18-35 years of age
* Free from musculoskeletal injury
* Do not participate in more than 4 hour of vigorous exercise per week
* Not taking dietary supplement or pre workout supplements for at least 1 month prior to study start
* Can abstain from other exercise for the duration of damage part of the study (4 days)
* Willing to participate and adhere to the study protocol
* Willing to limit berry and/or cherry intake to one portion per day
* Not to change their dietary / workout habits throughout the study (apart from abstaining from exercise during the damage part of the study)
* Able to understand the participant information, health screening questionnaire and the informed consent information
* Willing to participate and sign the informed consent form

Exclusion Criteria:

* BMI ≥30
* Taking any medication that might affect the outcome of the study, such as anti-inflammatory and immunosuppressant drugs
* Performance enhancing drugs and recreational drugs
* Orthopedic problems that include muscle tears that might affect ability to perform exercise
* Subject has a significant history or current presence of treated or untreated cardiometabolic, gastrointestinal, bleeding disorder, diabetes mellitus, high blood pressure (BP) [systolic BP> 140 and/or diastolic BP> 90], thyroid disease, tachyarrhythmia, heart disease, kidney disease, or liver disease.
* Subject currently suffers from a sleep disorder and/or has a known history of (or is currently being treated for) clinical depression, eating disorder(s) or any other psychiatric condition(s), which in the opinion of the investigator, might put the subject at risk and/or confound the results of the study.
* Have a recent history of surgery that might affect physical performance
* Current smoker
* Significant recent or planned change in dietary habit
* Have lost more than 6 kg in the past 6 months or planning to lose weight in the next month
* Allergy to berries
* Drinking more than 2 alcoholic beverages per day on average in a week (total 14 units)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 41 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Muscle strength | baseline, 24, 48 and 72 hours post exercise
  Muscle strength will be measured via maximal isometric voluntary contractions (MIVCs) performed using a portable strain gauge (MIE Medical Research Ltd., Leeds, UK). The peak value from 3 maximal contractions (separated by 60 seconds) will be used for analysis.

SECONDARY OUTCOMES:
Change in passive muscle soreness | baseline, 24, 48 and 72 hours post exercise
  Passive muscle soreness will be reported on a 0-200 mm visual analogue pain scale with 0mm representing no pain at all and 200mm representing unbearably painful.
Change in limb girth | baseline, 24, 48 and 72 hours post exercise
  Limb girth will be measured at the mid-thigh to examine limb swelling. This will be determined by identifying the midpoint between the inguinal crease and the superior border of the patella the right leg whilst the participant remained standing in anatomical zero. The location will be marked with permanent marker to ensure consistency on subsequent days.
Change in creatine kinase | baseline, 24, 48 and 72 hours post exercise
  A venous blood sample will then be taken to examine creatine kinase (CK) concentrations to provide evidence that muscle damage has occurred.
Change in counter movement jump height | baseline, 24, 48 and 72 hours post exercise
  A secondary measure of muscle strength loss and recovery will be evaluated via counter movement jumps (CMJ) with an optical system to measure jump height in cm. With hands on their hips, participants will descend into a ~90° squat and jump vertically with maximal effort. The average of 3 maximal jumps (separated by 30 seconds) will be used for analysis.
Change in 30m sprint time | baseline, 24, 48 and 72 hours post exercise
  Participants will complete a single maximal effort 30 m sprint where sprint time will be recorded. The sprint will be initiated from a line 30 cm behind the start line in order to prevent false triggering of the timing gates (Brower, Utah, USA).
Change in pain pressure threshold | baseline, 24, 48 and 72 hours post exercise
  Pain pressure threshold will be measured with a handheld algometer and on a 0-200 mm visual analogue pain scale with 0mm representing no pain at all and 200mm representing unbearably painful. Pain pressure threshold will be assessed whilst participant lay supine, a cylindrical flat headed probe of 1cm in diameter will be applied to a pre-determined site upon the muscle to a total pressure of 60 N with pressure being applied at a rate of 10N/second. The muscle site that will be used is the vastus lateralis. Once a pressure of 60 N is reached, the participants will be asked to point on the 0-200mm visual analogue scale their feeling of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbrai University, Newcastle upon Tyne, Tyne & Wear, United Kingdom